CLINICAL TRIAL: NCT07103239
Title: Feasibility and Acceptability of Three Component Intervention for the Heart Failure Care for Rural Dwelling Participants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephen Clarkson, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300015100; 1K23HL179489-01 (NIH)
Record Dates: First submitted 2025-07-25; First posted 2025-08-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video Based Visits (Experimental): Patients assigned to remote consultation will receive a video-based visit with the HF care team using the software platform of the PI's eMedicine division
  Interventions: Behavioral: Video Based Visits
- Remote Self-Care Education (Experimental): The intervention will be regular training at designated intervals vs self-guided education
  Interventions: Behavioral: Remote Self-Care Education
- Remote Patient Monitoring (Experimental): The devices include a mobile device, blood pressure cuff, and digital scale. The Remote Patient Monitoring team will call the consented participant over the phone to help with setup and use of the devices
  Interventions: Behavioral: Remote Patient Monitoring

INTERVENTIONS:
Behavioral: Video Based Visits — Video based visit with Heart Failure team
  Arms: Video Based Visits
Behavioral: Remote Self-Care Education — Self Guided Training
  Arms: Remote Self-Care Education
Behavioral: Remote Patient Monitoring — Participant will use home devices to monitor blood pressure and weight; Participant will then send results to RN educator
  Arms: Remote Patient Monitoring

SUMMARY:
The purpose of this research study is to determine if using remote blood pressure monitoring and video-based consultation is an effective way to help patients in rural communities better manage their heart failure.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Heart Failure
* English speaking
* primary residence in counties of interest

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 3 months
  Feasibility will be measured by recruitment rates (number screened vs. number enrolled), retention rates (percentage of participants that complete study), and participation metrics. We will aim to enroll at least 40% of the patients we approach for recruitment, and complete follow-up in at least 80% of all enrolled subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided